CLINICAL TRIAL: NCT01526876
Title: Effect of Clevidipine on Intracranial Pressure, Cerebral Blood Flow, Brain Tissue Oxygenation and Brain Cellular Metabolism in Severely Hypertensive Patients With Acute Brain Injury
Brief Title: The Effect of Clevidipine on Intracranial Pressure and Cerebral Perfusion Pressure (CCP) in Brain Injured Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Terminated by Sponsor
Sponsor: Columbia University (Other)
Collaborators: The Medicines Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAF4096
Record Dates: First submitted 2012-02-02; First posted 2012-02-06 (Estimated); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Hypertension
Keywords: Intracranial Pressure; Cerebral Perfusion Pressure; Clevidipine Butyrate
MeSH Terms: conditions — Hypertension | interventions — clevidipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm drug study (Experimental): The effect of systemic blood pressure reduction using Clevidipine on intracranial pressure (ICP) and cerebral perfusion pressure (CCP)
  Interventions: Drug: clevidipine butyrate

INTERVENTIONS:
Drug: clevidipine butyrate — intravenous infusion dose range 1.0 mg/hr - 32 mg/hr titrate to blood pressure effect duration of infusion: 6 hours
  Other Names: Cleviprex

SUMMARY:
Patients with acute brain injury are at risk for complications such as increased pressure in the brain (intracranial pressure (ICP)), decreased blood flow, bleeding, and brain swelling (cerebral edema). Several studies have suggested that high blood pressure is associated with a worsening outcome possibly due to an increased rate of continued bleeding or rebleeding, as well as increased brain swelling (cerebral edema). High systemic (body) blood pressure (SBP) may also increase the risk of ongoing bleeding. Therefore lowering the blood pressure (BP) is critical, as continued bleeding occurs most frequently in patients with high BP.

Clevidipine Butyrate (Cleviprex) is a new medication approved by the FDA for the treatment of acute high blood pressure (hypertension). Cleviprex is given through an intravenous line (IV) and has the benefit of being faster acting and easier to control adjustments than other drugs used to treat high BP. Patients who have an acute brain injury and who have severe high BP may benefit from this faster acting medication.

For this study, eligible patients, 18 yrs of age or older, will have been admitted to the Neurocritical care unit within 24 hours after their brain injury, who have high systemic (body) SBP. The treating physicians will have already had multimodality brain monitoring placed for clinical management of the patient (standard care).

The investigators will use Cleviprex to lower their SBP and record brain pressure and brain blood flow measurements from the multimodality monitoring. Due to the severity of their brain injury most of the patients eligible for the study will be unable to provide consent. Informed consent will be sought from a surrogate (family member, spouse or close friend) according to Columbia University Medical Center guidelines.

Cleviprex is fast acting and effects are seen in about 90 seconds. The medication will be started at a low rate, and if the SBP still needs lowering, the dose increased every 90 seconds until the maximum FDA approved dose is reached. If the SBP is still high, another medication used to treat high blood pressure will be added (Cardene or labetolol).

Once the SBP is lowered and is stable, the Cleviprex will be continued for 6 hours. As part of standard care, patients have their blood pressure monitored continuously. After 6 hours the treating physician will make a determination to continue clinical management with cleviprex or another antihypertensive medication.

DETAILED DESCRIPTION:
This is an open-label, single arm, single center study in patients with hypertension in the setting of an acute brain injury. Approximately 15 patients admitted to the Columbia University Neurocritical Care Unit with intracerebral hemorrhage, subarachnoid hemorrhage or traumatic brain injury who are hypertensive and have neuromonitoring probes placed in the course of standard clinical management will be enrolled over a 10-12 month period. Patients must be hypertensive (SBP > 180mmHg), or have an elevated cerebral perfusion pressure (CPP) above 100 mm Hg and the decision has been made by the ICU team to initiate an infusion of clevidipine to maintain CPP within a target range of 70-90 mm Hg and SBP between 120-180mmHg.

Due to the decreased level of consciousness from their injury, the majority of patients will be unable to provide consent. Informed consent will be sought from a surrogate according to Columbia University Medical Center (CUMC) guidelines (See section 8-Informed Consent Process).

Clevidipine infusion will be used to treat hypertension within the first 24 hours after injury. Multi-modality brain monitoring will have been placed as standard care.

Clevidipine will be infused at an initial rate of 2.0 mg/h for the first 90 seconds and titrated to effect (CPP target range of 70-90 mm Hg) by either doubling or reducing the dose by 50% every 90 seconds (with dose ranging 0-32mg/h of continuous IV infusion).

At the end of 6 hours clevidipine treatment, the treating physician will make a determination to continue clinical management with clevidipine or change to another antihypertensive medication.

Patients will be monitored at 24 hours after infusion for liver function, triglycerides and lipase.

ELIGIBILITY:
Inclusion Criteria:

1. Coma (Glasgow Coma Scale (GCS) less than or equal to 8) due to any cause
2. Male and Female patients > 18 years.
3. Mechanically ventilated
4. Functional multimodality neuromonitoring bundle (intracranial pressure (ICP) monitor, Hemedex, Licox, and microdialysis) placed in the course of routine clinical management
5. Patient is hypertensive at the time of enrollment (CPP >100 mm Hg and/or SBP >180mmHg) and the decision has been made to start clevidipine butyrate in order to maintain CPP within 70-90 mm Hg and/or SBP <180mmHg
6. Patient has a minimum of 60 min of baseline brain multimodality monitoring prior to initiation of clevidipine -

Exclusion Criteria:

1. Absence of negative pregnancy test in women of child-bearing potential.
2. FiO2 >50%
3. Unable to maintain stable sedative infusion rates for 4 hours
4. Unable to maintain stable ventilator setting for 4 hours
5. Unable to maintain stable insulin infusion rates for 4 hours
6. Patient is currently receiving nicardipine infusion
7. Allergy to soybean oil or lecithin
8. Participation in other clinical research studies involving the evaluation of other investigational drugs or devices within 30 days of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-11; Primary Completion 2012-11 (Actual); Study Completion 2012-12-19 (Actual)

PRIMARY OUTCOMES:
Reduction in blood pressure | Up to 24 hours from the start of clevidipine infusion
  Systemic Blood Pressure will be monitored every minute for the first 30 mins, at 45 and 6 mins and then hourly for 6 hours of treatment. ICP will be monitored every 5 minutes from start of infusion up to 6 hours of treatment

SECONDARY OUTCOMES:
"Time to target" (below the CCP threshold and Percent time within the target CCP range) | Up to 24 hours from the start of infusion
  Will be looking at the "Time to target" (below the CCP threshold and Percent time within the target CCP range) to assess whether clevidipine is safe and effective for rapidly controlling blood pressure to achieve desired cerebral perfusion pressure (CCP).

CONTACTS AND LOCATIONS:
Overall Officials: Stephan A Mayer, MD, Principal Investigator — Columbia University